CLINICAL TRIAL: NCT01489267
Title: The Safety and Efficacy of Umbilical Cord Mesenchymal Stem Cells Transplantation in Hereditary Cerebellar Ataxia Patients
Brief Title: A New Method to Treat Hereditary Cerebellar Ataxia - Umbilical Cord Mesenchymal Stem Cells Transplantation
Acronym: SCA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: General Hospital of Chinese Armed Police Forces (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20111031SCA; 20111031limin (Other: neuralstemcell)
Record Dates: First submitted 2011-10-30; First posted 2011-12-09 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Hereditary Cerebellar Ataxia.
Keywords: cerebellar ataxia; hereditary disease; stem cell
MeSH Terms: conditions — Spinocerebellar Degenerations; Cerebellar Ataxia; Genetic Diseases, Inborn | interventions — Stem Cell Transplantation; Cell- and Tissue-Based Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): Ten patients in the group only receive nerve functional evaluation and electrophysiology examination before and 1,3,6,12 months after recruit. They will not accept cell therapy.
- Stem cell transplantation (Experimental): 10 patients in the group accept stem cell transplantation.
  Interventions: Other: stem cell transplantation

INTERVENTIONS:
Other: stem cell transplantation — The patients accepted 4 times stem cell transplantations through lumbar puncture, the time is 3-5days between two treatments and the dose is about 2 ml(including 1×10'7 cells).
  Other Names: Cell therapy.
  Arms: Stem cell transplantation

SUMMARY:
Hereditary cerebellar ataxia is a type of autosomal dominant genetic disease, lesions mainly involving the cerebellum, but the spinal cord and cranial nerves may also be some involvement. A total of 20 molecularly diagnosed SCA1 patients divided in two groups. One group accepted for the treatment of stem cell transplantation,the other group will be the control. Purpose of this project to prove that allogeneic umbilical cord mesenchymal stem cells are applied to clinical safely, and in the treatment of hereditary cerebellar ataxia is valid.

DETAILED DESCRIPTION:
After admission the patients accepted transplantation would receive physical examination, blood and urine tests, electrocardiogram, electrophysiologic study;evaluation of SCA1 symptoms (balance, walking, dexterity, tremor, memory, mood and concentration),then stem cell therapy：after stem cell prepared, the patients accepted 4 times stem cell transplantations through lumbar puncture, the time is 3-5days between two treatments. The control only receive evaluation of SCA1 symptoms .

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years of age
2. Molecularly diagnosed SCA1

Exclusion Criteria:

1. Cognitively impaired individuals
2. Schizophrenics
3. Patients with severe kidney and liver disease, epilepsy, heart disease, pulmonary disease, cardiac arrhythmia, diabetes insipidus, leukemia and some other central neural disease (such as Parkinson disease, accidence of brain vascular et al)
4. Age less than 18 years, age greater than 65 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
blood test | within one week before transplantation
  white blood cell、neutrophilic granulocyte、leukomonocyte；glutamic pyruvic transaminase(GPT)、glutamic oxalacetic transaminase、lactate dehydrogenase(LDH)、;hydroxybutyrate dehydrogenase(HBDH)、phosphocreatine kinase(CK)；acidum uricum(UA)、creatinine(Cr)、α1- microglobulin、β2- microglobulin；lymphotoxin(LCT). Tumor markers(AFP,CEA,CA125,CA15-3,CA19-9,CA72-4CY21-1,NSE) ,Lymphocytes classification
Nerve functional evaluation | within one week before transplantation
  1. Timed-up-and-go test ,5 minutes down-and-up test
  2. ICARS score
  3. Modified Falls Efficacy Scale
  4. Berg balance assessment
  5. Tremor Rating Scale:
     * Part A - Tremor location/severity rating
     * Part B -Handwriting and drawings
     * Part C - Functional disabilities resulting from tremor
  6. Questionnaires related to sleep, depression (Beck Depression Inventory) (BDI), alertness (Computerized Continuous Performing Tasks) and memory (Mini Mental State Examination)
blood test | 1 month after transplantation
  white blood cell、neutrophilic granulocyte、leukomonocyte；glutamic pyruvic transaminase(GPT)、glutamic oxalacetic transaminase、lactate dehydrogenase(LDH)、;hydroxybutyrate dehydrogenase(HBDH)、phosphocreatine kinase(CK)；acidum uricum(UA)、creatinine(Cr)、α1- microglobulin、β2- microglobulin；lymphotoxin(LCT). Tumor markers(AFP,CEA,CA125,CA15-3,CA19-9,CA72-4CY21-1,NSE) ,Lymphocytes classification
blood test | 3 months after transplantation
  white blood cell、neutrophilic granulocyte、leukomonocyte；glutamic pyruvic transaminase(GPT)、glutamic oxalacetic transaminase、lactate dehydrogenase(LDH)、;hydroxybutyrate dehydrogenase(HBDH)、phosphocreatine kinase(CK)；acidum uricum(UA)、creatinine(Cr)、α1- microglobulin、β2- microglobulin；lymphotoxin(LCT). Tumor markers(AFP,CEA,CA125,CA15-3,CA19-9,CA72-4CY21-1,NSE) ,Lymphocytes classification
blood test | 6 months after transplantation
  white blood cell、neutrophilic granulocyte、leukomonocyte；glutamic pyruvic transaminase(GPT)、glutamic oxalacetic transaminase、lactate dehydrogenase(LDH)、;hydroxybutyrate dehydrogenase(HBDH)、phosphocreatine kinase(CK)；acidum uricum(UA)、creatinine(Cr)、α1- microglobulin、β2- microglobulin；lymphotoxin(LCT). Tumor markers(AFP,CEA,CA125,CA15-3,CA19-9,CA72-4CY21-1,NSE) ,Lymphocytes classification
blood test | 12 months after transplantation
  white blood cell、neutrophilic granulocyte、leukomonocyte；glutamic pyruvic transaminase(GPT)、glutamic oxalacetic transaminase、lactate dehydrogenase(LDH)、;hydroxybutyrate dehydrogenase(HBDH)、phosphocreatine kinase(CK)；acidum uricum(UA)、creatinine(Cr)、α1- microglobulin、β2- microglobulin；lymphotoxin(LCT). Tumor markers(AFP,CEA,CA125,CA15-3,CA19-9,CA72-4CY21-1,NSE) ,Lymphocytes classification
Nerve functional evaluation | 1 month after transplantation
  1. Timed-up-and-go test ,5 minutes down-and-up test
  2. ICARS score
  3. Modified Falls Efficacy Scale
  4. Berg balance assessment
  5. Tremor Rating Scale:
     * Part A - Tremor location/severity rating
     * Part B -Handwriting and drawings
     * Part C - Functional disabilities resulting from tremor
  6. Questionnaires related to sleep, depression (Beck Depression Inventory) (BDI), alertness (Computerized Continuous Performing Tasks) and memory (Mini Mental State Examination)
Nerve functional evaluation | 3 months after transplantation
  1. Timed-up-and-go test ,5 minutes down-and-up test
  2. ICARS score
  3. Modified Falls Efficacy Scale
  4. Berg balance assessment
  5. Tremor Rating Scale:
     * Part A - Tremor location/severity rating
     * Part B -Handwriting and drawings
     * Part C - Functional disabilities resulting from tremor
  6. Questionnaires related to sleep, depression (Beck Depression Inventory) (BDI), alertness (Computerized Continuous Performing Tasks) and memory (Mini Mental State Examination)
Nerve functional evaluation | 6 months after transplantation
  1. Timed-up-and-go test ,5 minutes down-and-up test
  2. ICARS score
  3. Modified Falls Efficacy Scale
  4. Berg balance assessment
  5. Tremor Rating Scale:
     * Part A - Tremor location/severity rating
     * Part B -Handwriting and drawings
     * Part C - Functional disabilities resulting from tremor
  6. Questionnaires related to sleep, depression (Beck Depression Inventory) (BDI), alertness (Computerized Continuous Performing Tasks) and memory (Mini Mental State Examination)
Nerve functional evaluation | 12 months after transplantation
  1. Timed-up-and-go test ,5 minutes down-and-up test
  2. ICARS score
  3. Modified Falls Efficacy Scale
  4. Berg balance assessment
  5. Tremor Rating Scale:
     * Part A - Tremor location/severity rating
     * Part B -Handwriting and drawings
     * Part C - Functional disabilities resulting from tremor
  6. Questionnaires related to sleep, depression (Beck Depression Inventory) (BDI), alertness (Computerized Continuous Performing Tasks) and memory (Mini Mental State Examination)

SECONDARY OUTCOMES:
Urinal test | within one week before transplantation
  proteinum、akaryocyte、α1- microglobulin、β2- microglobulin
Electrophysiology examination | within one week before transplantation
  somatosensory evoked potential(SEP)、brain stem auditory evoked potential(BAEP)
Urinal test | 1 month after transplantation
  proteinum、akaryocyte、α1- microglobulin、β2- microglobulin
Urinal test | 3 months after transplantation
  proteinum、akaryocyte、α1- microglobulin、β2- microglobulin
Urinal test | 6 months after transplantation
  proteinum、akaryocyte、α1- microglobulin、β2- microglobulin
Urinal test | 12 months after transplantation
  proteinum、akaryocyte、α1- microglobulin、β2- microglobulin
Electrophysiology examination | 1 month after transplantation
  somatosensory evoked potential(SEP)、brain stem auditory evoked potential(BAEP)
Electrophysiology examination | 3 months after transplantation
  somatosensory evoked potential(SEP)、brain stem auditory evoked potential(BAEP)
Electrophysiology examination | 6 months after transplantation
  somatosensory evoked potential(SEP)、brain stem auditory evoked potential(BAEP)
Electrophysiology examination | 12 months after transplantation
  somatosensory evoked potential(SEP)、brain stem auditory evoked potential(BAEP)

CONTACTS AND LOCATIONS:
Overall Officials: Yihua An, doctor, Study Director — director of neural stem cell transplantation department in general hospital of chinese armed police forces
Locations (1):
- Yihua An, Beijing, China